CLINICAL TRIAL: NCT01330745
Title: Mesenteric Microcirculatory Function Study Through Sublingual Evaluation During Cardiopulmonary Bypass
Brief Title: Microcirculation in Cardiac Surgery
Acronym: MICROCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/121/HP
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Cardiac Disorder
Keywords: cardiopulmonary bypass; mesenteric; microcirculatory function
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aortic valve replacement (Other)
  Interventions: Other: sublingual microcirculatory evaluation

INTERVENTIONS:
Other: sublingual microcirculatory evaluation — TNF, ICAM, syndecan-1, heparan sulfate

SUMMARY:
The purpose of this study is to determine whether cardiopulmonary bypass affects mesenteric microcirculatory function, using sublingual evaluation, in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years old
* aortic valvular disease needing aortic valve replacement

Exclusion Criteria:

* Age<18 years old
* emergent cardiac surgery
* other cardiac surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Microcirculatory impairment | 36 months
  Mean flow index measurement and capillar density study

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Doguet, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France